CLINICAL TRIAL: NCT03482310
Title: Restoring High Dimensional Hand Function to Persons With Chronic High Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: A2654-R
Record Dates: First submitted 2018-03-16; First posted 2018-03-29 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injuries; Tetraplegia; Quadriplegia
Keywords: Brain computer interface; electric stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cortical Control of Grasp Patterns (Experimental): Participants will be asked to think about holding different shaped objects, and the recorded cortical signal patterns will be decoded to match those grasp shapes
  Interventions: Device: Using the Neuroport cortical recording array to determine the desired grasp pattern for a functional electrical stimulation (FES) system

INTERVENTIONS:
Device: Using the Neuroport cortical recording array to determine the desired grasp pattern for a functional electrical stimulation (FES) system — Participants will be asked to think about holding different shaped objects, and the recorded cortical signal patterns will be decoded to match those grasp shapes

SUMMARY:
This study is for people who have a paralyzed arm and hand from a spinal cord injury, who have also received a recording electrode array in the brain as part of the BrainGate study. The study will look at the ability of these participants to control different grasping patterns of the hand, both in virtual reality and in his/her actual hand. Movement of the participant's hand is controlled by a functional electrical stimulation (FES) system, which involves small electrodes implanted in the arm, shoulder and hand that use small electrical currents to activate the appropriate muscles.

DETAILED DESCRIPTION:
This work aims to advance Brain-Computer-Interfaces (BCls) to provide severely paralyzed persons a natural way of controlling Functional Electrical Stimulation (FES) neuroprostheses for restoring arm and dexterous hand movements. The prospect of using BCI technology for restoring arm and hand movements for reaching and grasping is based on the hypothesis that in a paralyzed human, there is a repeatable and understandable relationship between recordable brain activity and specific aspects of imagined arm movements. Many previous studies have attempted to understand the relationships between brain activity and arm and hand movements in able-bodied monkeys. Little is known about these same relationships in humans, and specifically within the context of trying to control an FES arm and complex hand system. This study will recruit persons who already have BCI and FES systems implanted to take advantage of the possibility of recording high resolution brain activity in human participants. Thus, from this study, we aim to gain a better understanding of how brain signals are related to specific aspects of arm and complex hand movements in humans with paralysis. Additionally, this study will test novel implementations of complex hand movement restoration in Veterans and other persons with chronic hand and arm paralysis.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively intact (able to follow instructions)
* A spinal cord injury resulting in at least partial arm paralysis
* Participant in BrainGate2 clinical trial, having already received an intracortical array and demonstrated the ability to use the neural signals to control a cursor on a monitor.

Exclusion Criteria:

* Profound visual impairments
* Participant in BrainGate2 clinical trial with insufficient recordable neural signals (such that the researchers cannot decode a movement intention command signal)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Ability to form appropriate grasp patterns | Through study completion, typically around 1 year
  The success rate for achieving a series of specified grasp patterns will be calculated. This will be a percentage of the target grasp patterns successfully achieved.

CONTACTS AND LOCATIONS:
Overall Officials: Abidemi B. Ajiboye, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data.

REFERENCES:
- See also: Home site of BrainGate clinical trial — https://www.braingate.org
- See also: Home site of ReHAB study — https://rehabstudy.org